CLINICAL TRIAL: NCT04805385
Title: Effects of Lactobacillus Plantarum PS128 in Patients With Tourette's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CMUH109-REC2-188
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Tourette's Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PS128 (Experimental): Subjects will consume the PS128 capsules every day, 2 capsules at a time, for 12 weeks.
  Interventions: Dietary Supplement: PS128
- Placebo (Placebo Comparator): Subjects will consume the placebo capsules every day, 2 capsules at a time, for 12 weeks.
  Interventions: Dietary Supplement: PS128
- Healthy Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: PS128 — Each PS128 capsule contained >1 × 10^10 colony forming units (CFU) with microcrystalline cellulose and weights 425 ± 25 mg The placebo capsules only contained 425 ± 25 mg microcrystalline cellulose
  Other Names: Placebo
  Arms: PS128; Placebo

SUMMARY:
To evaluate whether supplementing with PS128 can improve the symptoms and quality of life related to Tourette's disease in children.

DETAILED DESCRIPTION:
This is a randomized double-blind healthy control study and the implementation period is after Institutional Review Board (IRB) approval to December 31, 2023.

Experimental group: 80 subjects who meet the criteria for the admission of Tourette's disease will be enrolled. They will consume the PS128 or placebo capsules every day, 2 capsules at a time, for 12 weeks. Healthy control group: 40 subjects of the same age as the experimental group will be included, without any intervention measures, only collect stool sample once.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-18 years old
* Tourette's disease is diagnosed
* Make sure it is not caused by medication or other diseases
* Cause major interference in social interaction, study or work
* The healthy control group is not diagnosed with Tourette's disease, and is judged by PI

Exclusion Criteria:

* Have taken antibiotics within a month or are receiving antibiotic treatment
* Used probiotic products in powder, capsule or tablet form within two weeks (except yogurt, yogurt, Yakult and other related foods)
* Patients who have undergone hepatobiliary gastrointestinal surgery (except for colorectal polypectomy and appendectomy)
* Inflammatory bowel disease, such as Crohn's disease or ulcerative colitis
* Those with a history of cancer
* Those who are allergic to lactic acid bacteria products
* Those who are not suitable to participate judged by PI

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | From Baseline to 4, 8, and 12 Weeks Assessed
  The YGTSS scale refers to Yale Global Tic Severity Scale, and it is a rating tool used to gauge the course of Tourette's syndrome in patients.

SECONDARY OUTCOMES:
Beck Youth Inventories (BYI-II) | From Baseline to 12 Weeks Assessed
  The new Beck Youth Inventories™ Second Edition (BYI-2) uses five self-report inventories to assess symptoms of depression, anxiety, anger, disruptive behavior, and self-concept in children and adolescents.
Attention-Deficit/Hyperactivity Disorder Test (ADHDT) | From Baseline to 12 Weeks Assessed
  The test yields standard scores, percentile ranks, severity levels, and probability of ADHD.
Child Behavior Checklist (CBCL) | From Baseline to 12 Weeks Assessed
  The Child Behavior Checklist (CBCL) is a widely used caregiver report form identifying problem behavior in children. It is widely used in both research and clinical practice with youths.
Autism Behavior Checklist-Taiwan Version (ABCT) | From Baseline to 12 Weeks Assessed
  The Autism Behavior Checklist (ABC) is one component of the Autism Screening Instrument for Educational Planning (ASIEP) and is the only one that has been evaluated psychometrically. The ABC is a 57-item behavior rating scale assessing the behaviors and symptoms of autism for children 3 and older.
Visual Analogue Scale for GI symptoms (VAS-GI) | From Baseline to 12 Weeks Assessed
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in patients after taking PS128.
Gilles de la Tourette Syndrome-Quality of Life Scale (GTS-QOL) | From Baseline to 4, 8 and 12 Weeks Assessed
  The Gilles de la Tourette Syndrome-Quality of Life Scale (GTS-QOL) is a self-rated disease-specific questionnaire to assess health-related quality of life of subjects with GTS.
Gut microbiota | From Baseline to 12 Weeks Assessed
  Intestinal microbiota may contribute to the metabolic health of the human host and, when aberrant, to the pathogenesis of various common metabolic disorders including obesity, type 2 diabetes, non-alcoholic liver disease, cardio-metabolic diseases and malnutrition.
Clinical Global Impression Scale (CGI) | From Baseline to 4, 8 and 12 Weeks Assessed
  Clinical Global Impression Scale (CGI) severity item provided with a seven-point scale of severity of the patient's clinical condition (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients).
miRNA | From Baseline to 12 Weeks Assessed
  peripheral blood miRNA expressions

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided